CLINICAL TRIAL: NCT01572467
Title: DICER1 Mutations and miRNA in Ovarian and Testicular Sex Cord Stromal Tumors of Childhood
Brief Title: Studying Genes in Samples From Younger Patients With Ovarian or Testicular Sex Cord Stromal Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARAR12B2; COG-ARAR12B2 (Other: Children's Oncology Group); NCI-2012-00721 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARAR12B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2012-04-05; First posted 2012-04-06 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Childhood Germ Cell Tumor; Leydig Cell Tumor; Ovarian Cancer
Keywords: Leydig cell tumor; ovarian stromal cancer; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor
MeSH Terms: conditions — Leydig Cell Tumor; Ovarian Neoplasms; Testicular Neoplasms; Ovarian Germ Cell Cancer | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer.

PURPOSE: This research trial is studying genes in tumor samples from younger patients with ovarian or testicular sex cord stromal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the role of DICER1 mutations and miRNA pathways in the etiology and progression of ovarian or testicular sex cord stromal tumors.

OUTLINE: Archived tumor tissue samples are analyzed for D1CER1 mutation and mRNA expression by reverse-transcriptase polymerase chain reaction (RT-PCR) and laser micro dissector. Results are then correlated with medical data, including age at diagnosis, diagnosis, pathology report, presenting symptoms, family history, treatment, outcome, and length of follow-up, when available.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Fixed and frozen tissue samples from the ATBR01 B1 tissue bank and from the International Pleuropulmonary Blastoma Registry, Children's Hospital of Boston, and Massachusetts General Hospital
* Tissue samples from patients diagnosed with:

  * Ovarian

    * Sertoli-Leydig cell tumor
    * Juvenile granulosa cell tumor
    * Adult granulosa cell tumor
    * Gynandroblastoma
    * Sex cord stromal tumor with annular tubules
    * Sex cord stromal tumor, undifferentiated
    * Sertoli tumor
    * Leydig tumor
  * Testicular:

    * Granulosa cell tumor
    * Sertoli tumor
    * Leydig tumor
    * Sertoli-Leydig
    * Undifferentiated stromal tumor

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Ovarian or Testicular Sex Cord Stromal Tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Correlation between DICER1 mutations and miRNA pathways with outcomes using descriptive analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dana A. Hill, MD, Principal Investigator — Children's National Research Institute